CLINICAL TRIAL: NCT05289154
Title: Self- Applied Acupressure and Online Qigong for Patients Suffering From Chronic Fatigue After Corona Virus Infection 19 (COVID-19) - a Randomized Controlled Mixed-methods Study.
Brief Title: Acupressure and Qigong in Chronic Fatigue Post COVID-19.
Acronym: ACUQiG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACUQiG
Record Dates: First submitted 2022-03-18; First posted 2022-03-21 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Post-COVID-19 Syndrome
Keywords: post COVID-19, sequelae, chronic fatigue
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Naturopathy

STUDY DESIGN:
Intervention Model Description: Prospective, randomised controlled, confirmatory intervention study with mixed methods approach
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self- applied acupressure plus Qigong plus advice literature (Experimental): daily 20 min of self- applied acupressure over 8 weeks on acupuncture points Yintang, LI4, Pe6, ST36, SP6 and depending on further symptoms plus DU23/24 in hyposmia, LU7 in dyspnoea, GB34 in pain conditions, GB20 in headache OR Anmian in sleeping disorders.
  The 16 sessions of 45 min Qigong course over 8 weeks will contain live online guided exercises with breathing, stretching and tapping of meridians and exercises such as the crane exercise.
  Interventions: Other: self- applied acupressure plus Qigong course plus advice literature
- advice literature (Active Comparator): advice literature contains naturopathic remedies such as application of massage-oils, use of herbal teas, meditation techniques, breathing exercises for reconvalescence after COVID19.
  Interventions: Behavioral: advice literature with naturopathy

INTERVENTIONS:
Other: self- applied acupressure plus Qigong course plus advice literature — daily self applied acupressure over 20min plus 2 times per week online live Qigong course of each 45min- both over 8 weeks.
  Arms: self- applied acupressure plus Qigong plus advice literature
Behavioral: advice literature with naturopathy — advice literature with naturopathic remedies will be handed out and application will be supported with dairies and phone calls
  Arms: advice literature

SUMMARY:
International observational studies confirm the high incidence of post-infectious residual syndrome after infection with severe acute respiratory syndrome corona virus 2 (SARS-COV2), which can occur in 10-15% of all infected persons, regardless of the severity of the acute infection. Post corona virus disease 19 (postCOVID-19) patients suffer mostly from symptoms such as fatigue, muscle pain, problems to focus, depression and sleep disturbances.

So far, there are no results of interventional studies for the treatment of chronic fatigue post COVID-19, but there are indicators that post COVID-19 syndrome is a chronic subclinical inflammation, similar to Chronic Fatigue Syndrome / Myalgic Encephalomyelitis CSF/ME, which also often develops from a postviral syndrome. Previously tested and effective strategies for the treatment of chronic fatigue syndrome / myalgic encephalomyelitis (CFS/ME) will be tested in the treatment of chronic fatigue postCOVID-19, in this randomized controlled trial a combination of acupressure and Qigong.

The aim of this project is to evaluate an acupressure treatment plus a Qigong exercise series specifically tailored for chronic fatigue postCOVID-19 , used daily by the patients themselves and regularly supervised, in comparison to the advice literature on the treatment of PostCOVID-19 syndrome alone.

DETAILED DESCRIPTION:
Prospective two-arm (parallel groups) randomised controlled confirmatory intervention study with mixed methods approach in 2x 100 patients (n=200).

Intervention: self-applied acupressure and online Qigong course over 8 weeks and follow up at week 16.

Group 1: Acupressure + Qigong: Massage of the points daily for 3 minutes per point with the finger or an acupuncture pen (some points can be massaged bilaterally, therefore total approx. 20 min). In addition, twice a week an online guided Qigong course with a duration of 30-45 min. The patients should practise Qigong at least 3 times a week (including the course date). In addition, all patients will receive the guidebook literature for the treatment of complaints after SARS-CoV2 infection.

Group 2: Patients will receive advice literature on the treatment of chronic fatigue after SARS-CoV2 infection. After the end of this study the patients of this group will receive written information and video material regarding the acupressure and Qigong exercises.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of chronic fatigue (after SARS-CoV2 infection)
2. with at least 3 of 7 criteria at time of study inclusion: sleeping disorder, headaches, joint pain/muscle pain, anxiety/depression, memory impairment/ concentration problems, anosmia, exercise intolerance.
3. acute SARS-CoV2 infection at least 12 weeks ago
4. age 18-60 years
5. visual analogue scale (0-100 mm) physical resilience of maximum 60 mm
6. SF-36 physical function of maximum 65
7. technically equipped to participate in the online intervention and willing to follow the study procedure, acupressure and Qigong to perform the exercise series at home
8. written informed consent available.

Exclusion Criteria:

1. fatigue already present before the SARS-CoV2 infection
2. other underlying diseases leading to symptoms of chronic fatigue, such as major depression, oncological diseases, multiple sclerosis, fibromyalgia and drug abuse
3. other serious underlying diseases, such as severe pulmonary, cardiac, psychiatric or infectious diseases, which could interfere with study participation or affect the results
4. ongoing opioid therapy or opioid therapy in the week prior to study entry
5. chronic use of cannabinoids before or during the study.
6. start of psychotherapy or interruption of ongoing therapy during study participation
7. female participants: pregnancy or breastfeeding
8. participation in another clinical intervention study during study participation
9. ongoing pension procedure or planned claiming of a pension procedure due to disability
10. planned inpatient rehabilitation measures during study participation due to PostCOVID-19 -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 Physical Function subscale | week 8
  Primary study objective is to assess the changes in the mean score of the SF-36 Physical Function subscale between the two study arms assessing the degree of fatigue.

SECONDARY OUTCOMES:
EQ5D (EuroQoL 5 domains) | week 8 and 16
  disease specific QoL
SF36 PFS (Short Form 36 physical function subscale) | week 16
  changes in the mean score of the SF-36 Physical Function subscale- assessing the degree of fatigue
Chalder Fatigue-Scale | week 8 and 16
  Fatigue severity
VAS physical resilience (visual analogue scale) | week 8 and 16
  visual analogue scale for subjective physical resilience
PHQ9 (Patient Health Questionnaire 9) | week 8 and 16
  Patient Health Questionnaire assessing depression
VAS pain (visual analogue scale) | week 8 and 16
  visual analogue scale for subjective pain
hand grip strength | week 8 and 16
  hand grip strength
Spirometry | week 8 and 16
  forced expiratory volume
autonomic dysfunction orthostasis test | week 8 and 16
  heart rate and blood pressure analysis in orthostasis
d2- test | week 8 and 16
  test for concentration- ability to focus
qualitative substudy | week 8 and 16
  interviews regarding experience of illness and therapy

CONTACTS AND LOCATIONS:
Overall Officials: Benno Brinkhaus, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold DT, Hamilton FW, Milne A, Morley AJ, Viner J, Attwood M, Noel A, Gunning S, Hatrick J, Hamilton S, Elvers KT, Hyams C, Bibby A, Moran E, Adamali HI, Dodd JW, Maskell NA, Barratt SL. Patient outcomes after hospitalisation with COVID-19 and implications for follow-up: results from a prospective UK cohort. Thorax. 2021 Apr;76(4):399-401. doi: 10.1136/thoraxjnl-2020-216086. Epub 2020 Dec 3. PMID 33273026
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Chan JSM, Ng SM, Yuen LP, Chan CLW. Qigong exercise for chronic fatigue syndrome. Int Rev Neurobiol. 2019;147:121-153. doi: 10.1016/bs.irn.2019.08.002. PMID 31607352
- [Background] Jason L, Brown M, Evans M, Anderson V, Lerch A, Brown A, Hunnell J, Porter N. Measuring substantial reductions in functioning in patients with chronic fatigue syndrome. Disabil Rehabil. 2011;33(7):589-98. doi: 10.3109/09638288.2010.503256. Epub 2010 Jul 9. PMID 20617920
- [Background] Glasier CM, Seibert JJ, Williamson SL, Seibert RW, Corbitt SL, Rodgers AB, Lange TA. High resolution ultrasound characterization of soft tissue masses in children. Pediatr Radiol. 1987;17(3):233-7. doi: 10.1007/BF02388167. PMID 3295732
- [Background] Weyand CM, Goronzy JJ. The role of infectious agents in the etiopathogenesis of chronic rheumatic diseases. Verh Dtsch Ges Inn Med. 1990;96:319-24. doi: 10.1007/978-3-642-84317-4_58. No abstract available. PMID 2092449
- [Derived] Bauer T, Grabowska W, Ortiz M, Bellmann-Strobl J, Engelhardt U, Nogel R, Hummelsberger J, Michalsen A, Roll S, Stockigt B, Batram H, Mietzner A, Scheibenbogen C, Willich SN, Paul F, Brinkhaus B, Dietzel J. Self-medication and off-label prescribing in post COVID-19 syndrome: Baseline data of a randomized acupressure and qigong trial. Integr Med Res. 2025 Sep;14(3):101197. doi: 10.1016/j.imr.2025.101197. Epub 2025 Jul 5. PMID 40727709